CLINICAL TRIAL: NCT02499068
Title: Proyecto Madrileño Sobre el Manejo de la Enfermedad Pulmonar Obstructiva Crónica Con Telemonitorización a Domicilio. (Multicentre Project on the Home Telemonitoring of Patients With Severe Chronic Obstructive Pulmonary Disease).
Brief Title: Madrid Project on the Management of Chronic Obstructive Pulmonary Disease With Home Telemonitoring
Acronym: PROMETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arturo Garcia (Other)
Collaborators: Linde Health Care (Other); Técnicas Avanzadas de Investigación en Servicios de Salud TAISS (Unknown); Syreon Corporation (Industry)
Responsible Party: Sponsor-Investigator, Arturo Garcia, Fundación Teófilo Hernando, Fundación Teófilo Hernando, Spain
Organization: Fundación Teófilo Hernando, Spain (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROMETE
Record Dates: First submitted 2015-03-20; First posted 2015-07-15 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: COPD; Disease Progression
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- COPD, Telehealth (Experimental): Patients randomized to this arm would be followed by home telehealth devices and monitored on a daily bases for early detection of exacerbations and prompt clinical intervention.
  Interventions: Device: Telehealth
- COPD, Normal clinical practice (No Intervention): Patients would do the usual clinical practice.

INTERVENTIONS:
Device: Telehealth — Monitoring devices installed at patients home and patients are monitored on a daily bases for early detection of exacerbations and prompt clinical intervention.and being follow-up on a daily bases for early detection and prompt intervention.
  Other Names: Telemedicine
  Arms: COPD, Telehealth

SUMMARY:
The purpose of the study is to verify the clinical effectiveness of a managed home telemonitoring program in patients with severe COPD against usual clinical practice, as measured by the decrease in the number of exacerbations, number of hospitalizations, hospital days and emergency room visits in a 12 month period

The primary endpoint of effectiveness is "severe exacerbations avoided."

The main hypothesis is that patients with severe or very severe COPD patients managed with a home telehealth program have better outcomes than patients managed according to usual clinical practice.

DETAILED DESCRIPTION:
Randomized, controlled, multicenter, performance, cost assessment and economic evaluation clinical trial. An arm of the trial will consist of patients assigned to the intervention group (telehealth group: TG ), and the other arm will consist of patients randomized to the control group (routine clinical practice: RCP).

For the economic evaluation, the perspective of the health system will be used. Therefore it only direct costs will be considered. In the TG arm also intervention costs it will be considered.

Patient selection:

Responsible researcher at each hospital center will coordinate the patient selection process. The researchers will identify candidate patients screening through hospital medical records.

After this first screening, patients will be contacted and invited to participate in the study. In a personal interview, the researcher explains the study to the patient and deliver the information sheet, verifying that patient meets all inclusion/exclusion criteria, obtains informed consent and then proceeds to patient randomization. To avoid bias from exclusions, researchers will hold record with patient exclusion causes.

Every hospital centers will include on average 60 patients (30 in each arm). The inclusion of patients will be competitive; having centers including patients in the study until reaching the final sample size of 120 patients per arm.

Randomization:

To avoid selection bias, patients assigned to each group will be randomized. To ensure that the number of subjects in each arm is the same, a restrictive block randomization is performed. Randomization is performed using random number generation by computer and the block size of 10 units.

Home Telehealth program:

Vital sign devices being used: spirometer, pulse oximeter with capacity for heart rate monitor, blood pressure, Visionox® (device capable of measuring respiratory rate, compliance with the hours of oxygen, and the flow and pattern of oxygen used).

Devices send data automatically to a modem by Bluetooth. Modem receives and transmits data simultaneously from the monitoring devices to a Central Monitoring Center (CMC). Data received by the modem are encrypted and sent to the telehealth monitoring platform via a 3G signal.

The CMC is manned by registered nurses and operates during office hours, 7 days a week.

Nurses will attend the patient's home for: the installation of the telehealth devices; to perform a thorough training of the patients / caregivers in the use of equipment and the COPD telehealth program.

Patients will perform daily vital sign measurements at the same time, at rest, after administration of the medication and the pattern of oxygen used. Visionox® performs measurements of respiratory rate and oxygen adherence automatically.

Measured data will be monitored on a daily bases by the nurses at the CMC. CMC will follow-up information, filter for fle positives and false negatives, and use an application acting as a traffic light system:

* Green: meant that measurements had been taken and were within the predefined limits, and no further action was required.
* Yellow: "technical alert". This means that the measurements had not been taken or had not been received. This alert could lead to a "clinical alert" due to a lack of adherence or discouragement. When the parameters were not received the nurse at the CMC called the patient to find the reason behind the alert, and either ruled out medical causes or, if one, notified the researcher leading the study.
* Red: "clinical alert". Meant that a measurement exceeded the limits that were previously preestablished for each.

Classification of severity of clinical alerts is performed by the CMC according to an algorithm. Depending n severity different early medical interventions are taken, or escalated to clinical responsible for early intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being over 50 and under 90 years of age.
* Being diagnosed with COPD according to the criteria of GesEPOC, with severe airflow obstruction defined as a forced expiratory volume in one second (FEV1) less than 50% of theoretical.
* "Exacerbator phenotype" defined as COPD patients having two or more moderate or severe exacerbations per year (GesEPOC guide). These exacerbations should be separated by at least 4 weeks after the end of previous treatment or 6 weeks from the start in cases that have not been treated
* Clinically stable condition, defined as 6 weeks without clinical symptoms since the last exacerbation of COPD.
* Having home oxygen therapy.
* Sign the informed consent.

Exclusion Criteria:

* Inability of the patient or caregiver to understand the procedure of Telehealth program.
* Have a life expectancy of less than one year.
* Have terminal heart failure (NYHA functional class III-IV).
* Having advanced renal insufficiency (creatinine clearance <30%) or be on dialysis program.
* Have liver cirrhosis or be included in a program of liver transplantation.
* Be institutionalized or in Residential hospice care.
* Having a mini-mental test-score less than 24, because this score suggests dementia
* To be considered by your doctor as not comply the treatment or monitoring required by their lung disease.
* Failure to meet any of the inclusion criteria.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Number of hospitalizations due to exacerbation of COPD avoided | 1 year

SECONDARY OUTCOMES:
Cost-efficiency of treatment | 1 year
Cost-utility of treatment | 1 year
satisfaction of both patients and clinician responsibility questionnaire | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Julio Ancochea Bermúdez, MD, PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (5):
- Spain (5):
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Rey Juan Carlos, Madrid

REFERENCES:
- [Background] Segrelles Calvo G, Gomez-Suarez C, Soriano JB, Zamora E, Gonzalez-Gamarra A, Gonzalez-Bejar M, Jordan A, Tadeo E, Sebastian A, Fernandez G, Ancochea J. A home telehealth program for patients with severe COPD: the PROMETE study. Respir Med. 2014 Mar;108(3):453-62. doi: 10.1016/j.rmed.2013.12.003. Epub 2013 Dec 16. PMID 24433744
- [Derived] Ancochea J, Garcia-Rio F, Vazquez-Espinosa E, Hernando-Sanz A, Lopez-Yepes L, Galera-Martinez R, Peces-Barba G, Perez-Warnisher MT, Segrelles-Calvo G, Zamarro C, Gonzalez-Ponce P, Ramos MI, Conforto JI, Jafri S, Soriano JB. Efficacy and costs of telehealth for the management of COPD: the PROMETE II trial. Eur Respir J. 2018 May 30;51(5):1800354. doi: 10.1183/13993003.00354-2018. Print 2018 May. No abstract available. PMID 29599185